CLINICAL TRIAL: NCT04755244
Title: A Phase 1/2 Study of Evorpacept (ALX148) in Combination With Venetoclax and Azacitidine in Patients With Acute Myeloid Leukemia (AML) (ASPEN-05)
Brief Title: A Study of Evorpacept (ALX148) With Venetoclax and Azacitidine for Acute Myeloid Leukemia (ASPEN-05)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: While intended to be a Phase 1/2 clinical study, the study never moved forward to Phase 2.
Sponsor: ALX Oncology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT148005
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2023-08

CONDITIONS: Acute Myeloid Leukemia; AML, Adult
Keywords: ALX148; CD47; SIRPalpha; azacitidine; venetoclax; evorpacept
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ALX148; venetoclax; Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- evorpacept (ALX148) + venetoclax + azacitidine (Experimental): Phase 1a: Participants will receive escalating doses of evorpacept (ALX148) in combination with venetoclax and azacitidine
  Phase 1b/2: Participants will receive evorpacept (ALX148) at the recommended Phase 2 dose in combination with venetoclax and azacitidine.
  Interventions: Drug: evorpacept; Drug: venetoclax; Drug: azacitidine

INTERVENTIONS:
Drug: evorpacept — Fusion protein that blocks CD47-SIRPalpha pathway
  Other Names: ALX148
Drug: venetoclax — BCL-2 inhibitor
  Other Names: Venclexta
Drug: azacitidine — Hypomethylating agent (HMA)
  Other Names: Vidaza

SUMMARY:
This Phase 1/2 clinical study will evaluate evorpacept (ALX148) in combination with venetoclax and azacitidine for the treatment of patients with acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
The Phase 1 will consist of a dose escalation of evorpacept (ALX148) in combination with venetoclax and azacitidine to evaluate safety and tolerability, and to identify the recommended Phase 2 dose of evorpacept (ALX148) in combination with venetoclax and azacitidine. The Phase 2 will evaluate the efficacy of evorpacept (ALX148) in combination with venetoclax and azacitidine for patients with AML. While intended to be a Phase 1/2 clinical study, the study never moved forward to Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed diagnosis of relapsed/refractory or newly diagnosed AML per WHO 2016 classification.
* Phase 1a: AML that is relapsed/refractory or that is previously untreated in patients not considered suitable for intensive induction therapy.
* Phase 1b: AML that is relapsed/refractory after prior treatment with a HMA-based regimen.
* Phase 2: Previously untreated AML in patients who are not considered suitable candidates for intensive induction therapy.
* Adequate renal and liver function.
* Age ≥18 years.
* Adequate performance status.

Exclusion Criteria:

* In Phase 1a and 1b, patients that have undergone prior allo-HSCT must be at least 3 months post-HSCT, without uncontrolled graft-versus-host disease (GVHD). For Phase 2, patients that have undergone prior allo-HSCT are excluded.
* Patients with newly diagnosed AML with favorable risk cytogenetics such as t(8;21), inv(16), or t(16;16) as per the NCCN Guidelines Version 3, 2019 for AML.
* Patients with acute promyelocytic leukemia (APL).
* Prior treatment with any anti-CD47 or anti-SIRPalpha (signal regulatory protein alpha) agent.
* Known active viral infections, including hepatitis B and C, human immunodeficiency virus (HIV), acquired immunodeficiency syndrome (AIDS) related illness, or SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Phase 1: Dose Limiting Toxicities (DLT) | Up to 28 days
  Number of participants with a DLT
Phase 2: Composite complete remission rate (CRc) | Approximately 6 months
  Number of participants achieving a complete remission (CR) and complete remission with incomplete hematologic recovery (CRi) per European LeukemiaNet (ELN) 2017 criteria

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marks JA, Wang X, Fenu EM, Bagg A, Lai C. TP53 in AML and MDS: The new (old) kid on the block. Blood Rev. 2023 Jul;60:101055. doi: 10.1016/j.blre.2023.101055. Epub 2023 Feb 14. PMID 36841672